

Statistical Analysis Plan (SAP) for Study UB-313-101

A First-in-Human Study to Evaluate the Safety, Tolerability, and Immunogenicity of UBITh® Migraine Immunotherapeutic Vaccine (UB-313) in Healthy Participants

Date: 7 November 2023

Version 2.0



## Signature Page

I have reviewed this Statistical Analysis Plan and approve its contents.

| Author<br>Study Statistician | Signature: Date: 11/9/2023 |
|---|---|
| Project Statistician | Signature: Date: 11/9/2023 |
| Senior Director, Clinical Development<br>Global Product Lead<br>Vaxxinity, Inc. | Signature:<br>Date: 11/9/2023 |
| Director, Clinical Operations<br>Vaxxinity, Inc. | Signature: Date: 11/9/2023 |



#### **Contents**

| Signature | e Page | 2 |
|------------|------------------------------------------------------------|----|
| 1.0 | Introduction | |
| 2.0 | Study Objectives and Design | 4 |
| 2.1 | Objectives and Endpoints | 4 |
| 2.2 | Study Design | 6 |
| 3.0 | Analysis Sets | 7 |
| 4.0 | General Consideration | 7 |
| 5.0 | Statistical Analyses | 8 |
| 5.1 | Immunogenicity, Pharmacodynamics, and Exploratory Analyses | 8 |
| 5.1.1 | Immunogenicity Analyses | 8 |
| 5.1.2 | Pharmacodynamics (PD) Analyses | 10 |
| 5.1.3 | Other Exploratory Analyses | 12 |
| 5.2 | Safety Analyses | 12 |
| 5.2.1 | Extent of Exposure | 13 |
| 5.2.2 | Treatment Tolerability | 13 |
| 5.2.3 | Adverse Events | 13 |
| 5.2.4 | Laboratory Data | 15 |
| 5.2.5 | Other Safety Parameters | 16 |
| 5.3 | Other Analyses | 16 |
| 5.3.1 | Study Participants | 16 |
| 6.0 | Additional details not mentioned in the protocol | 18 |
| 7.0 | Version History | 18 |
| List of Ta | ables | |
| Table 1. | Objectives and Endpoints | 5 |
| List of Ap | ppendices | |
| Appendix 1 | List of Abbreviations | 19 |
| Appendix 2 | MedDRA Terms for AESI | 21 |



#### 1.0 Introduction

This Statistical Analysis Plan (SAP) provides describes the statistical analyses outlined and specified in the Protocol UB-313-101 Version 2.0: A First-in-Human Study to Evaluate the Safety, Tolerability, and Immunogenicity of UBITh® Migraine Immunotherapeutic Vaccine (UB-313) in Healthy Participants, dated 14 June 2022.

#### 2.0 Study Objectives and Design

#### 2.1 Objectives and Endpoints

The primary, secondary, and exploratory objectives and endpoints of this study are shown below.



**Table 1. Objectives and Endpoints** 

| Objectives | Endpoints |
|---|---|
| <b>Primary Safety and Tolerability</b> | |
| To evaluate the safety and tolerability of UB-313, when administered at selected dose regimens given intramuscularly (IM) to healthy adults. | Safety will be assessed by adverse events (AEs), adverse events of special interest (AESIs), medically attended adverse events (MAAEs), local (injection site) and systemic (generalized) reactions (i.e., reactogenicity), clinical laboratory assessments (e.g., chemistry, hematology, urinalysis), vital signs, neurological and physical examinations and electrocardiograms (ECGs), through the end of study. |
| Primary Immunogenicity | |
| To evaluate the anti-Calcitonin Gene-Related Peptide (anti-CGRP) specific antibody responses to selected UB-313 dose regimens in healthy adults. | Immunogenicity will be measured serum anti-CGRP antibody titers and analyzed from baseline to Week 16 and Week 44. |
| Secondary | |
| To evaluate the effects of selected UB-313 dose regimens on capsaicin-induced dermal blood flow (DBF) as a surrogate marker of target engagement. | Pharmacodynamics (PD) of the immune response will measured by the inhibition of capsaicin-induced increase in DBF and will be analyzed from baseline to Week 16 and until return to baseline or until Week 44, whichever comes first. |
| Exploratory | |
| To evaluate the effects of selected UB-313 dose regimens on CGRP concentrations in serum. | CGRP concentrations in serum through the end of study. |
| To characterize antibodies generated by UB-313. | Antibody titers against components of the UB-313 (i.e., CpG1 and UBITh1) through the end of study. Isotype-specific anti-CGRP antibody titers through the end of study. |



| To examine cytokine release induced by | Cytokine release from peripheral blood |
|---|---|
| UB-313. | mononuclear cell (PBMC)s stimulated with |
| | component of the UB-313 (T-cell ELISpot) |
| | through Week 16. |

#### 2.2 Study Design

This is a single-site, randomized, double-blind, placebo-controlled, multi-dose regimen, first-in-human study of UB313, an anti-CGRP peptide-based immunotherapy candidate. Details for study design are described in protocol section 3.

The study design is shown in

Figure 1.

**Figure 1 Study Design Schematic** 



<sup>\*</sup>No more than 4 participants will be dosed in a 24-hour period.

Abbreviations: C (capsaicin Challenge); EoS (End of Study); EoT (End of Treatment); M (month); SCR (Screening Period); h (hour); Wk (week).

<sup>\*</sup>No more than 4 participants will be dosed in a 24-hour period.



SRC (Safety Review Committee) is responsible for the safety review and dose escalation decision. At the end of Week 16, an EoT analysis will be performed for each cohort, unblinded by treatment cohort and pooled by dose on all safety, tolerability, immunogenicity and DBF data. At the end of the treatment analysis, study team members who are responsible for the conduct and data management of the study, and participants will remind blinded to the subject level treatment assignment. If there are no safety concerns, the study will continue until all participants complete Week 44 (End of Study [EoS]) visit. An unblinded statistics team from an external CRO (AvanSight) will perform the EOT and EOS analyses.

#### 3.0 Analysis Sets

The following populations sets will be used for the analyses.

- Full Analysis Set (FAS) consists of all participants randomized and received all three administrations of study Investigational Medicinal Product (IMP) per protocol, and who have at least one evaluable post baseline assessment of the anti-CGRP antibody titers.
- Safety Analysis Set (SS) consists of all participants who receive at least 1 dose of study IMP.

Demographic, baseline, and safety analysis will be based on Safety Analysis Set. Immunogenicity analyses, pharmacodynamics (PD) analyses, and exploratory analyses will be performed for FAS.

#### 4.0 General Consideration

All analyses will be conducted using observed data only and no missing data will be imputed.

In general, the baseline value is defined as the last available value before the first injection of study dose.

All analysis and summary will be performed by dose group, defined as below:

- 100/100/100µg (8 active participants in cohort 1)
- 300/100/100µg (8 active participants in cohort 2)



- 300/300/300µg (8 active participants in cohort 3)
- 600/100/100µg (8 active participants in cohort 4)
- Placebo (8 participants from all cohorts)

#### 5.0 Statistical Analyses

# 5.1 Immunogenicity, Pharmacodynamics, and Exploratory Analyses

Efficacy analysis will be based on FAS. All analyses and plot will be performed by dose group for each visit and each timepoint unless otherwise specified. In general, summary of a variable (e.g., titer, CIDBF) will include baseline, actual value, and change (or percent change) from baseline when applicable. Summary plots will be done when applicable.

For qualtititive assessements (e.g., titer value, CIDBF...), the distribution will be examined. If the distribution is similar to log normal, log transformation will be applied. In this case, geometric mean and GMR (Geometric Mean Ratio) will be presented in place of mean and difference. For model analysis, log transformed value will be used, analysis results will be presented after anti log transformation.

#### 5.1.1 Immunogenicity Analyses

## 5.1.1.1 Serum anti-CGRP Antibody Titers (Primary Endpoint and Analysis)

The primary immunogenicity endpoint is serum anti-CGRP antibody titers.

The anti-CGRP antibody titers and change from baseline will be summarized at each visit.

Comparison between each UB-313 groups and Placebo group in change from baseline will be based on an analysis of covariance (ANCOVA) model including dependent variable of change from baseline in titer values at each postbaseline visit, with factor of treatment, and baseline titer as covariate.



## 5.1.1.2 Serum anti-CGRP Antibody Titers vs Age and Gender (Exploratory)

Relationship between immunogenicity and age, and gender differences in immunogenicity will be explored.

Serum anti-CGRP antibody titers will be summarized by gender.

#### 5.1.1.3 Seroconversion and Responder Rate (Exploratory)

Additional exploratory endpoints are seroconversion status and sero responder status for each participant.

Seroconversion is defined as the ratio (i.e., geometric mean fold change) of post baseline titer over baseline titer  $\geq X$  (e.g., X=1, 2, 3, 4).

Seroconversion rates will be calculated for all postbaseline visits along with 95% CIs based on Binomial distribution. In addition, the difference in the response rates between UB-313 and the placebo group (UB-313 – placebo) will be calculated, and the 95% CIs based on Fisher's Exact test will be displayed.

To define the threshold of response, mean and standard deviation of titer values will be calculated using the assessments below.

- Titer values at baseline from all participants and
- Titer values at all postbaseline visits up to Week 16 from placebo participants.

The mean plus two standard deviations (mean+2SD) will be used as the threshold of response. Responders will be defined as the participants with titer value greater than or equal to response threshold for each visit including baseline and postbaseline visits.

Responder analysis will be done similarly to seroconversion rates.

# 5.1.1.4 Cumulative AUC for Serum anti-CGRP Antibody Titer and C<sub>max</sub> (Exploratory)

Cumulative AUC is defined as the area under the curve from Day 1 to each scheduled visit. AUC will be calculated by the sum of individual trapezoid area under the curve of level of antibodies.



AUC from baseline to each postbaseline visit will be calculated. AUC above baseline for each postbaseline will also be calculated (i.e., derive AUC using each postbaseline value change from baseline). In the case of early dropout, the AUC will be calculated up to the last visit with titer values. AUC will not be calculated for the visits after dropout.

 $C_{max}$  is the highest observed value up to end of study (EoS).  $C_{max}$  change from baseline will be calculated as  $C_{max}$  – baseline value.

ANCOVA model will include dependent variable of cumulative AUC and AUC above baseline, with factor of dose group, and baseline titer as covariate.  $C_{max}$  and  $C_{max}$  change from baseline will be analyzed similarly.

#### 5.1.1.5 Quantitative anti-CGRP Antibody Titers (Exploratory)

Quantitive anti-CGRP antibody titers will be summrized.

#### 5.1.2 Pharmacodynamics (PD) Analyses

## 5.1.2.1 Capsaicin Induced Dermal Blood Flow (Secondary Endpoint and Analysis)

#### Capsaicin-induced increase in DBF (CIDBF)

The pharmacodynamics (PD) endpoint is the inhibition of capsaicin-induced increase in DBF (CIDBF). The DBF at each timepoint at each visit will be calculated as the average of two capsaicin-induced locations.

The DBF will be summarized for each timepoint (i.e., 0, 15, 30, 45, and 60 minutes) at each visit (i.e., Day 1, Day 29, Day 57, Day 85, Day 113, and Day 141, Day 197, Day 253, Day 309 as applicable).

#### Change and Percent Change from pre capsaicin in CIDBF

For each post capsaicin time point at each visit, change and percent change from pre capsaicin will be calculated. For example, change at 30 minutes post capsaicin on Day 29 from pre capsaicin is calculated as the DBF at 30 minutes post capsaicin on Day 29 minus the DBF at 0-minute pre capsaicin on Day 29. Percent change will be calculated similarly.



Summary will be presented. Between dose group comparison will be done. ANCOVA model will include dependent variable of change (or percent change) from pre capsaicin in CIDBF, with factor of dose group, and DBF at 0-minute pre capsaicin as covariate.

#### Change and Percent Change from Baseline (Day 1 prior to study IMP) in CIDBF

For 30 minutes and 45 minutes post capsaicin at each visit, change and percent change from baseline (Day 1 prior to study IMP) will be calculated. For example, change from baseline at 30 minutes post capsaicin on Day 29 is calculated as the DBF at 30 minutes post capsaicin on Day 29 minus the DBF at 30 minutes post capsaicin on Day 1 prior to study IMP. Percent change will be calculated similarly.

Summary will be presented. Between dose group comparison will be done. ANCOVA model will include dependent variable of change (or percent change) from baseline in CIDBF, with factor of dose group, and DBF at baseline (Day 1 prior to study IMP) as covariate.

#### DBF for Non-capsaicin Vehicle Control

DBF from control location (vehicle RD) will be summarized for each dose group and each visit as well as for pooled group and all visits.

#### 5.1.2.2 CIDBF by Gender (Exploratory)

DBF and change from pre capsaicin will be summarized by gender for baseline, week 16 and week 44.

#### 5.1.2.3 CIDBF AUC (Exploratory)

CIDBF AUC (0-60min) and change from baseline (<u>Day 1 prior to study IMP</u>) will be summarized by dose group for each visit. Between dose group comparison will be done. ANCOVA model will include dependent variable of AUC, with factor of dose group, and baseline AUC as covariate.

#### 5.1.2.4 Inhibition Responder (Exploratory)

CIDBF at 30 minutes post capsaicin will be used for the responder analysis. To define threshold of response, mean and standard deviation will be calculated using the assessments below.

• CIDBF at baseline from all participants



The mean minus two standard deviations (mean-2SD) will be used as the threshold of response. CIDBF responders will be defined as the participants with CIDBF less than or equal to response threshold for each visit including baseline and postbaseline visits.

Responder analysis will be done similarly to seroconversion rates.

#### 5.1.2.5 Duration of Inhibition Response (Exploratory)

Duration of inhibition response is defined as from baseline to either return to baseline or until Week 44, whichever comes first for inhibition responders. Participants who do not return to baseline will be censored at the time of study exit.

Duration of inhibition response will be summarized for each dose group, using Kaplan-Meier product-limit estimates.

#### 5.1.3 Other Exploratory Analyses

#### 5.1.3.1 CGRP Concentrations in Serum

Summary will be done.

## 5.1.3.2 Correlation between CIDBF, anti-CGRP Antibody, aCGRP Concentrations

Correlation between CIDBF AUC (0 to 60 minutes) and anti-CGRP antibody at each visit will be summarized separately by dose group. Pearson's corelation coefficient will be calcaluated.

In addition, correlation between CIDBF AUC (0 to 60 minutes) and aCGRP concentrations, aCGRP concentrations and anti-CGRP antibody at each visit will be done similarly.

#### 5.1.3.3 Antibodies Against Components of UB-313

Antibody titers against components of UB-313 (include but are not limited to anti-CGRP target epitope, anti-UBITh, and anti-CpG1) will be summarized.



#### 5.1.3.4 Cytokine Release included by UB-313

# 5.2 Cytokine release from peripheral blood mononuclear cell (PBMC)s stimulated with component of UB-313 (T-cell ELISpot) will be summarized.Safety Analyses

Safety will be assessed by Adverse Events (AEs), Adverse Event of Special Interests (AESIs), medically attended adverse events (MAAEs), local (injection site) and systemic (generalized) reactions (i.e., reactogenicity), clinical laboratory assessments, vital signs, physical neurological and examinations and electrocardiograms (ECGs), through the end of study. Safety analysis will be based on safety analysis set.

#### 5.2.1 Extent of Exposure

The number of injections and total dosage of study drug will be summarized.

#### 5.2.2 Treatment Tolerability

Overall treatment tolerability will be summarized in the safety population.

The overall treatment tolerability of UB-313 for each dose group is defined as the percentage of number of administered doses divided by number of administered doses plus number of missed doses of participant(s) who drops out due to drug-related AE(s). It is calculated according to the following formula:

$$100\% \text{ x } (A+B1+C+D) / (A+B1+B2+C+D)$$

where

A: number of administered doses of completers

B1: number of administered doses of participant(s) who drops out due to drug-related AE(s)

B2: number of missed doses of participant(s) who drops out due to drug-related AE(s)

C: number of administered doses of participant(s) who drops out due to drug-unrelated AE(s)

D: number of administered doses of participant(s) who drops out not due to AE(s)



#### 5.2.3 Adverse Events

Adverse events (AEs) will be coded using MedDRA. The actual version of MedDRA will be noted in the statistical tables and clinical study report. The intensity of the AEs is graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

An AE will be considered a treatment-emergent adverse event (TEAE) if the AE began or worsened (increased in severity or became serious) after the first administration of study drug.

A treatment-emergent serious adverse event (TESAE) is defined as an SAE that is also a TEAE.

TEAEs will be summarized by participant incidence rates. The number and percentage of participants with TEAEs will be tabulated for overall (i.e., any preferred term), as well as by primary MedDRA SOC and PT.

#### 5.2.3.1 Adverse Event Overview

An overview of AEs will be presented. The number and percentage of participants experiencing at least one event will be summarized for each of the below categories.

- Treatment related TEAE
- Serious TEAE
- Treatment related serious TEAE
- Adverse events of special interest (AESI)
   AESI is defined in Protocol Appendix 4 ADVERSE EVENTS OF INTEREST.
   AESI MedDRA terms based on Protocol Table 5 AESIs based on identified adverse reactions and Table 6 AESIs based on important potential risks are listed in Appendix 2.
- Medically attended adverse event (MAAE)
- Death

#### 5.2.3.2 Treatment-Emergent Adverse Events

The number and percentage of participants will be tabulated for the below categories of TEAEs.

- TEAEs by SOC and PT
- TEAEs by SOC, PT and maximum severity



- TEAEs by SOC, PT and maximum relationship
- Treatment-related TEAEs by SOC and PT
- SAEs (including deaths) by SOC and PT
- TEAEs leading to treatment discontinuation by SOC and PT
- AESIs by SOC and PT
- MAAEs by SOC and PT

#### 5.2.3.3 Solicited Adverse Events

Solicited local and systemic AEs are defined in protocol section 7.5.3.2 Reactogenicity Assessment, and protocol appendix 3: Toxicity grading scale for solicited adverse events.

Local (injection site) and systemic (generalized) reactions (i.e., reactogenicity) after each study product injection will be presented by maximum severity. Summary will include counts and percentages of participants by dose group for each reaction and each injection.

#### 5.2.4 Laboratory Data

#### 5.2.4.1 Hematology and Chemistry Parameters

Clinical laboratory values will be reported in International System of Units (SI) units and categorized based on normal ranges collected from laboratories.

Summary and plot will be presented.

The number and percentage of participants who experienced laboratory test abnormalities will be summarized for each lab assay.

For each scheduled postbaseline visit, shift from baseline will be presented based on the categories below:

- Low, Clinically Significant
- Low, Not Clinically Significant
- Normal
- High, Not Clinically Significant
- High, Clinically Significant

Unscheduled visits will be presented in listings but will not be included in summaries.



#### 5.2.4.2 Other Laboratory Parameters

Quantitative data for all other laboratory parameters will be presented using descriptive statistics of values and absolute changes from baseline to each visit. Shift tables will be presented when applicable.

Other laboratory parameters include urinalysis, inflammatory markers, cytokine panel (The cytokine panel will include but is not limited to IFN- $\gamma$ , IL-2, IL-4, IL-6, IL-8, and TNF- $\alpha$ ).

#### 5.2.4.3 Vital Signs

Descriptive statistics for semi-recumbent vital signs including heart rate (HR), systolic and diastolic blood pressure (BP), respiratory rate (RR), body temperature at each visit will be presented.

#### 5.2.4.4 Neurological Examinations

Results will be summarized or listed.

#### 5.2.4.5 Physical Examinations

Results will be summarized or listed.

#### 5.2.4.6 Electrocardiograms (ECGs)

Descriptive statistics for triplicate ECG parameters and changes from baseline values at each visit will be presented. Shift from baseline to the worst postbaseline will be presented.

#### 5.2.5 Other Safety Parameters

#### 5.2.5.1 Height and Weight

Descriptive summary will be done.

#### 5.2.5.2 Pregnancy Test

Positive results will be listed.



5.3 Other Analyses

#### 5.3.1 Study Participants

#### 5.3.1.1 Disposition of Participants

The total number of participants will be summarized below.

• Participants who were screened (who signed informed consent)

Number and percentage of participants in each of the following categories will be summarized.

- Participants who were randomized (this is denominator for the percentages described below
- Participants who received at least one dose of study drug
- Participants who completed treatment period (Week 16)
- Participants who discontinued during the treatment period
  - o Reasons for treatment discontinuation (based on reasons reported on CRF)
- Participants who completed the study
- Participants who discontinued from the study
  - o Reasons for study discontinuation (based on reasons reported on CRF)

Number of participants in each analysis population will be summarized. Participants excluded from analysis will be listed.

In addition, reasons for screen failure will be summarized.

#### 5.3.1.2 Protocol Deviations

Major protocol deviations will be summarized.

#### **5.3.1.3** Demographics and other Baseline Characteristics

#### 5.3.1.3.1 Demographics

Demographic parameters (age, gender, race, and ethnicity) will be summarized.

#### 5.3.1.3.2 Baseline characteristics

Baseline parameters (height, body weight, BMI) will be summarized.



#### 5.3.1.4 Medical History

Medical history and surgical history that are not ongoing at the trial initiation, and medical history that are ongoing at the trial initiation will be summarized separately. The number and percentage of participants will be tabulated by MedDRA SOC and PT. The actual version of MedDRA will be noted in the statistical tables and clinical study report.

#### **5.3.1.5** Prior and Concomitant Medications

A prior medication is defined as any medication taken prior to the start of study treatment. A concomitant medication is defined as any medication taken after the start of study treatment (i.e., any medication that started prior to the study treatment and continued to be taken after the study treatment or any medication that started after the study treatment).

Prior and concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary. The actual version of WHO will be noted in the statistical tables and clinical study report. The number and percentage of participants reporting prior or concomitant medications will be summarized separately by Anatomical Therapeutic Chemical (ATC) 1st level class and preferred drug name. If more than one medication is coded to the same preferred drug name for the same participant, the participant will be counted only once for that preferred drug name.

#### 6.0 Additional details not mentioned in the protocol

Additional details and specifications have been included in this SAP to allow for better understanding of the intended methods. Additional analyses (including exploratory and subgroup assessments) for select variables have been added. Additional sensitivity analyses will be conducted to explore any effects related to the presence of data outliers.

#### 7.0 Version History

| SAP<br>Version | Approval<br>Date | Change | Rationale |
|----------------|------------------|----------------|------------------|
| 1 | 17 May 2023 | Not Applicable | Original version |



| 2 | Added AUC above baseline for anti-CGRP antibody titers in section 5.1.1.4. | To adjust for baseline. |
|---|---|---|
| | Added C <sub>max</sub> for anti-CGRP antibody titers in section 5.1.1.4. | To capture maximum titer level. |
| | Added text for CI DBF AUC in section 5.1.2.3. | Updated for clarity. |
| | Moved cytokine release from section 5.2.4.2 to section 5.1.3.4. | Updated for clarity. |



## **Appendix 1 List of Abbreviations**

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| ADA | Anti-drug antibody |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ANCOVA | Analysis of Covariance |
| BP | Blood pressure |
| CI | Confidence interval |
| COVID-19 | Coronavirus disease 2019 |
| CRF | Case report form (electronic or paper) |
| CRO | Contract research organization |
| DBP | Diastolic blood pressure |
| ECG | Electrocardiogram |
| EOS | End of study |
| EOT | End of treatment |
| FIH | First-in-human |
| GMR | Geometric Mean Ratio |
| HR | Heart rate |
| IMP | Investigational Medicinal Product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NA | Not applicable |
| NCS | Not clinically significant |
| PE | Physical examination |
| PD | Pharmacodynamic |
| PP | Pulse pressure |
| PT | Preferred term |
| SAE | Serious adverse event |



| Abbreviation | Definition |
|--------------|----------------------------------|
| SS | Safety analysis set |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| VS | Vital signs |



## Appendix 2 MedDRA Terms for AESI

| | | Primary System Organ | |
|---|---|---|---|
| Preferred Term Code | Preferred Term | Class Code | Primary System Organ Class |
| 10047340 | Vertigo | 10013993 | Ear and labyrinth disorders |
| 10010774 | Constipation | 10017947 | Gastrointestinal disorders |
| 10028034 | Mouth ulceration | 10017947 | Gastrointestinal disorders |
| 10030985 | Oral mucosa bleeding | 10017947 | Gastrointestinal disorders |
| 10042128 | Stomatitis | 10017947 | Gastrointestinal disorders |
| 10016256 | Fatigue | 10018065 | General disorders and administration site conditions |
| 10022052 | Injection site bruising | 10018065 | General disorders and administration site conditions |
| 10022061 | Injection site erythema | 10018065 | General disorders and administration site conditions |
| 10022075 | Injection site induration | 10018065 | General disorders and administration site conditions |
| 10022086 | Injection site pain | 10018065 | General disorders and administration site conditions |
| 10022093 | Injection site pruritus | 10018065 | General disorders and administration site conditions |
| 10022094 | Injection site rash | 10018065 | General disorders and administration site conditions |
| 10022095 | Injection site reaction | 10018065 | General disorders and administration site conditions |
| 10053425 | Injection site swelling | 10018065 | General disorders and administration site conditions |
| 10030095 | Oedema | 10018065 | General disorders and administration site conditions |
| 10042674 | Swelling | 10018065 | General disorders and administration site conditions |
| 10002198 | Anaphylactic reaction | 10021428 | Immune system disorders |
| 10002218 | Anaphylaxis | 10021428 | Immune system disorders |
| 10020751 | Hypersensitivity | 10021428 | Immune system disorders |
| 10028810 | Nasopharyngitis | 10021881 | Infections and infestations |
| 10028334 | Muscle spasms | 10028395 | Musculoskeletal and connective tissue disorders |
| 10001760 | Alopecia | 10040785 | Skin and subcutaneous tissue disorders |
| 10002424 | Angioedema | 10040785 | Skin and subcutaneous tissue disorders |
| 10005191 | Blister | 10040785 | Skin and subcutaneous tissue disorders |
| 10064579 | Exfoliative rash | 10040785 | Skin and subcutaneous tissue disorders |
| 10037087 | Pruritus | 10040785 | Skin and subcutaneous tissue disorders |
| 10037844 | Rash | 10040785 | Skin and subcutaneous tissue disorders |
| 10037855 | Rash erythematous | 10040785 | Skin and subcutaneous tissue disorders |
| 10037876 | Rash papular | 10040785 | Skin and subcutaneous tissue disorders |
| 10037884 | Rash pruritic | 10040785 | Skin and subcutaneous tissue disorders |
| 10046735 | Urticaria | 10040785 | Skin and subcutaneous tissue disorders |

#### Certificate Of Completion

Envelope Id: 614EBD33C7E04C5A9BE3B7D924AD5905

Subject: Complete with DocuSign: Vaxxinity UB-313-101 SAP v2.0\_7Nov2023\_clean.pdf

Source Envelope:

Document Pages: 22 Certificate Pages: 5

Signatures: 4 Initials: 0

AutoNav: Enabled

**Envelopeld Stamping: Enabled** 

Time Zone: (UTC-08:00) Pacific Time (US & Canada)

Status: Completed

**Envelope Originator:** 

505 Odyssey Way Mailbox 204 Vaxxinity Merritt Island, FL 32953 @vaxxinity.com

IP Address: 204.197.150.156

#### Record Tracking

Status: Original

11/9/2023 11:41:50 AM

Holder:

Location: DocuSign

#### Signer Events

@vaxxinity.com

Associate Director, Clinical Operations Security Level: Email, Account Authentication (None)

Signature

Timestamp

Sent: 11/9/2023 11:43:50 AM Viewed: 11/9/2023 12:15:38 PM Signed: 11/9/2023 12:16:02 PM

#### **Electronic Record and Signature Disclosure:**

Accepted: 11/9/2023 12:15:38 PM ID: 98a255eb-0679-408d-90ea-298da57f4f37

(None)

Sr. Director, Clinical Development

Security Level: Email, Account Authentication (None)

@vaxxinity.com

**Electronic Record and Signature Disclosure:** 

Using IP Address:

Signature Adoption: Drawn on Device

Using IP Address:

@vaxxinity.com

Signature Adoption: Pre-selected Style

Signed using mobile

Sent: 11/9/2023 11:43:50 AM Viewed: 11/9/2023 12:14:53 PM Signed: 11/9/2023 12:15:06 PM

Accepted: 6/29/2022 6:51:02 AM

ID: 86667a7c-4adb-4b39-a43c-3caee5c4b247

Using IP Address:

Signature Adoption: Pre-selected Style

Sent: 11/9/2023 11:43:50 AM Viewed: 11/9/2023 12:07:16 PM Signed: 11/9/2023 12:07:26 PM

Security Level: Email, Account Authentication

**Electronic Record and Signature Disclosure:** 

ID: 86369ec0-4b7b-44ac-96eb-7dc5220a2924

Accepted: 11/13/2022 2:06:40 PM

Security Level: Email, Account Authentication (None)

Signature Adoption: Pre-selected Style Using IP Address:

#### **Electronic Record and Signature Disclosure:**

Accepted: 11/9/2023 12:07:48 PM ID: a201a6dc-2d3c-49ac-8637-f6836601a00c Sent: 11/9/2023 11:43:51 AM Viewed: 11/9/2023 12:07:48 PM Signed: 11/9/2023 12:08:22 PM

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete | Hashed/Encrypted<br>Security Checked | 11/9/2023 11:43:51 AM<br>11/9/2023 12:07:48 PM |
| Completed | Security Checked<br>Security Checked | 11/9/2023 12:08:22 PM<br>11/9/2023 12:16:02 PM |
| | - | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Vaxxinity Inc. - Non Regulated (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### How to contact Vaxxinity Inc. - Non Regulated:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: it@vaxxinity.com

#### To advise Vaxxinity Inc. - Non Regulated of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at it@vaxxinity.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Vaxxinity Inc. - Non Regulated

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to it@vaxxinity.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Vaxxinity Inc. - Non Regulated

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to it@vaxxinity.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Vaxxinity Inc. Non Regulated as described above, you
  consent to receive exclusively through electronic means all notices, disclosures,
  authorizations, acknowledgements, and other documents that are required to be provided
  or made available to you by Vaxxinity Inc. Non Regulated during the course of your
  relationship with Vaxxinity Inc. Non Regulated.